CLINICAL TRIAL: NCT04210778
Title: Combined Model of Online Remote Interventions for Cancer-Related Cognitive Impairment
Acronym: CRCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Israel cancer research fund (Unknown); Israel Cancer Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRCI-HMO-CTIL
Record Dates: First submitted 2019-12-01; First posted 2019-12-26 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Cognitive Decline; Cancer
Keywords: Cancer related cognitive impairment; Telerehabilitation; Computerized Cognitive training; Adult cancer survivors; Functional treatment
MeSH Terms: conditions — Cognitive Dysfunction; Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trail (RCT)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomization will take place only after the investigator will complete baseline assessment, so the assessment procedure wont be affected by group allocation. In addition, the investigator who will assess the outcomes post intervention and at 3 month follow up will be blind to the intervention allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CRAFT (Cognitive Training and Functional Treatment) (Experimental): Over 12 weeks this group will be instructed to complete 3 weekly sessions of Computerized Cognitive Training, in addition to a weekly 1 hour remote CO- OP (Meta cognitive strategy training) session. Each participant will set three occupational goals that will be the focus of the CO -OP treatment
  Interventions: Behavioral: Cognitive orientation to daily occupational performance (CO-OP); Behavioral: Computerized Cognitive Training (BrainHQ, posit science)
- Computerized Cognitive Training (Active Comparator): This group will be instructed to complete 3 weekly sessions of Computerized Cognitive Training
  Interventions: Behavioral: Computerized Cognitive Training (BrainHQ, posit science)
- Treatment As Usual (No Intervention): This group will receive no intervention

INTERVENTIONS:
Behavioral: Cognitive orientation to daily occupational performance (CO-OP) — The CO-OP is a client-centered, goal directed approach aimed at enabling individuals to identify strategies that will improve daily function. A Weekly (1hr) session is delivered remotely via video conferencing.
  Arms: CRAFT (Cognitive Training and Functional Treatment)
Behavioral: Computerized Cognitive Training (BrainHQ, posit science) — The BrainHQ training targets multiple cognitive domains. The training will be delivered remotely, using a web-based program. Training progresses in an adaptive, individualized manner, based on individual progression of each participant . Participants are required to practice a minimum of half hour, three times a week (total of 1.5hr)
  Arms: CRAFT (Cognitive Training and Functional Treatment); Computerized Cognitive Training

SUMMARY:
Cancer survival rates have increased dramatically in recent years. However, many survivors report cognitive decline following treatment, which significantly impairs their quality of life. Online cognitive training programs have shown promise in improving cognitive functions in cancer survivors, but most studies report limited impact of training on everyday function. A complementary treatment approach is functional treatment delivered by occupational therapists, which directly targets daily function. Combining the two approaches has the potential to overcome the limitations of both approaches, enabling improved cognitive functions and transfer to daily function. Remotely-administrated interventions further make treatment accessible and cost-effective. The current study is aimed at testing the efficacy of a novel, combined, remotely-delivered treatment approach: Cognitive Retraining and Functional Treatment(CRAFT), using a Randomized Controlled Trial (RCT) design. 90 cancer survivors will be randomly assigned to receive 15 weeks of either the combined treatment, computerized training only, or treatment-as-usual. Outcomes will be assessed at completion, and following 3 months of no contact, to test immediate and enduring effects of treatment. Baseline predictors for treatment response will be further assessed.

Positive results in the proposed study could potentially change the therapeutic landscape for rehabilitation of cancer-related cognitive decline, which currently impair the lives of millions worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18;
2. Subjective concern about declines in cognitive functioning related to a diagnosis of cancer and/or cancer related treatment. This will be obtained by asking participants the question "do you have concerns about your memory or other thinking abilities following cancer treatment?". Participants are required to answer yes to this question.
3. interested in treatment and state they have 2 weekly hours available for the intervention.
4. Completion of active treatment for non-Central Nervous System (CNS) cancer (e.g., chemotherapy,radiation therapy and surgery) 6 months or more in the past.
5. Cognitive decline with no dementia: 21<Mini-Mental State Examination <27 (Folstein, Folstein, & McHugh, 1975) and/or 19< Montreal Cognitive Assessment <26 (Nasreddine et al., 2005);
6. Daily access to a computer and Internet facilities;
7. Able to sign an informed consent;
8. Stable psychiatric condition (according to participants self- report and medical file).

Exclusion Criteria:

1. no prior experience using computers;
2. pregnancy;
3. History of a central nervous system tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change in the Canadian Occupational Performance Measure (COPM) (Law et al., 1998) | Time 0: Baseline, before group allocation and intervention; Time 1: at completion of intervention, an average of 15 weeks after T0; Time 2: 3 months after Time 1 (an average of 6 months after enrollment)
  A semi-structured interview used to assess the self-perception of clients' performance and satisfaction with their level of participation in daily functioning regarding the five most important problems they identified. The patient rates each problem on a 10-point scale indicating his level of performance (1= not able to do it at all, 10= able to do it extremely well) and level of satisfaction (1= not satisfied at all, 10 = extremely satisfied). Change is assessed by administering the interview at different time points.
Change in Computerized Cognitive Assessments (Posit Science) | Time 0: Baseline, before group allocation and intervention; Time 1: at completion of intervention, an average of 15 weeks after T0; Time 2: 3 months after Time 1 (an average of 6 months after enrollment)
  Computerized Assessment will be used to assess neuro-cognitive function using five different tasks from posit science. Domains that will be assessed are sustained attention, visual working memory, speed of processing (visual and auditory) and flexibility
Change in Functional Assessment of Cancer Therapy - Cognition (FACT COG) (Jacobs, Jacobsen, Booth-Jones, Wagner, & Anasetti, 2007) | Time 0: Baseline, before group allocation and intervention; Time 1: at completion of intervention, an average of 15 weeks after T0; Time 2: 3 months after Time 1 (an average of 6 months after enrollment)
  A self-report questionnaire for cancer patients with cognitive function issues. The tool includes 37-items assessing memory, concentration, language and thinking abilities. The items are grouped into 4 subscales: perceived cognitive impairment (PCI), perceived cognitive abilities (PCA), comments from others (OTH), and impact on quality of life (QOL). The items are rated on a 5-point Likert scale (0=never, 4 =several times a day) regarding the past 7 days, higher scores indicating greater QOL.

SECONDARY OUTCOMES:
Change in the Functional Assessment of Cancer Therapy-General practice (FACT-GP) (Cella et al., 1993) | Time 0: Baseline, before group allocation and intervention; Time 1: at completion of intervention, an average of 15 weeks after T0; Time 2: 3 months after Time 1 (an average of 6 months after enrollment)
  A patient reported quality of life questionnaire commonly used in cancer survivors. The tool consists of 21-statements on which the respondent is asked to think of the last week and determine his level of agreement to each statement on a 5-point scale (0=not at all, 4= very strongly agree), higher scores indicate greater QOL.
Change in the Patient Health Questionnaire (PHQ-9)(Kroenke, Spitzer, & Williams, 2001) | Time 0: Baseline, before group allocation and intervention; Time 1: at completion of intervention, an average of 15 weeks after T0; Time 2: 3 months after Time 1 (an average of 6 months after enrollment)
  A self-report measure for the screening and severity of depressive symptomatology. The nine items in the questionnaire regard the frequency of symptoms within the last 2 weeks and are rated on a four-point Likert scale (0= not at all, 3=almost every day). The maximum score is 27, with higher scores reflecting more depressive symptoms.
Change in the Generalized Anxiety Disorder (GAD -7) (Spitzer, Kroenke, Williams, & Löwe, 2006) | Time 0: Baseline, before group allocation and intervention; Time 1: at completion of intervention, an average of 15 weeks after T0; Time 2: 3 months after Time 1 (an average of 6 months after enrollment)
  A self-report measure used for the screening and severity of GAD, It includes 7 items describing the severity of the patient's anxiety over the past 2 weeks on a four- point Likert scale (0= not at all sure, 3= nearly every day). The sum score ranges from 0 to 21, with values of 5, 10, 15 indicated mild, moderate or severe anxiety symptoms
Change in the Ruminative Response Scale (RRS) (Treynor, Gonzalez, & Nolen-Hoeksema, 2003) | Time 0: Baseline, before group allocation and intervention; Time 1: at completion of intervention, an average of 15 weeks after T0; Time 2: 3 months after Time 1 (an average of 6 months after enrollment)
  A self-report questionnaire used to assess rumination among adults. The RRS includes 22 items describing responses to depressed mood. Items are rated on a 4-point Likert scale (1= almost never, 4= almost always). A total score can be calculated, summing all 22 items scores (22-88), higher scores indicating more rumination.
Change in the Functional Assessment of Cancer Therapy - Fatigue (FACT -F) (Yellen, Cella, Webster, Blendowski, & Kaplan, 1997) | Time 0: Baseline, before group allocation and intervention; Time 1: at completion of intervention, an average of 15 weeks after T0; Time 2: 3 months after Time 1 (an average of 6 months after enrollment)
  A fatigue measure used to assess cancer patients at the active or survivor stage. The 13-item questionnaire utilizing a five-point Likert scale (0 = not at all, 4=very much so). The total score varies from 0 - 52, higher score indicating more fatigue
Change in the New General Self-Efficacy Scale (NGSE) (Chen, Gully, & Eden, 2001) | Time 0: Baseline, before group allocation and intervention; Time 1: at completion of intervention, an average of 15 weeks after T0; Time 2: 3 months after Time 1 (an average of 6 months after enrollment)
  A self administered questionnaire used to evaluate self-efficacy. The questionnaire includes eight items that are rated on a five- point Likert scale (1= strongly disagree, 5=strongly agree). The total score ranges from 9 to 40, with higher scores reflecting better self-efficacy.
Change in Performance Quality Rating Scale (PQRS) (Martini, Rios, Polatajko, Wolf, & McEwen, 2015) | Time 0: Baseline, before group allocation and intervention; Time 1: at completion of intervention, an average of 15 weeks after T0; Time 2: 3 months after Time 1 (an average of 6 months after enrollment)
  An observational measure, used to assess actual performance of client-selected activities. Score ranges between 1 (0% task completion) to 10 (100% of task completion) and is established by therapist thoroughly questioning client about performance using explicit questions.
Social Presence (Hauber, Regenbrecht, Billinghurst, & Cockburn, 2006) | 3 Time points during intervention (Week 1, Week 5, Week 10), CRAFT only
  A questionnaire used to measure co-presence and social presence of adults participating in technology based social interactions
Satisfaction questionnaire and interview | Time 1: At completion of intervention (an average of 15 weeks after baseline) (CRAFT only)
  A satisfaction questionnaire and interview were developed for the use of this study

CONTACTS AND LOCATIONS:
Overall Officials: Yafit Gilboa, PhD, Principal Investigator — Hebrew University of Jerusalem
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Von Ah D, Carpenter JS, Saykin A, Monahan P, Wu J, Yu M, Rebok G, Ball K, Schneider B, Weaver M, Tallman E, Unverzagt F. Advanced cognitive training for breast cancer survivors: a randomized controlled trial. Breast Cancer Res Treat. 2012 Oct;135(3):799-809. doi: 10.1007/s10549-012-2210-6. Epub 2012 Aug 24. PMID 22918524
- [Background] Cicerone KD, Goldin Y, Ganci K, Rosenbaum A, Wethe JV, Langenbahn DM, Malec JF, Bergquist TF, Kingsley K, Nagele D, Trexler L, Fraas M, Bogdanova Y, Harley JP. Evidence-Based Cognitive Rehabilitation: Systematic Review of the Literature From 2009 Through 2014. Arch Phys Med Rehabil. 2019 Aug;100(8):1515-1533. doi: 10.1016/j.apmr.2019.02.011. Epub 2019 Mar 26. PMID 30926291
- [Background] Lange M, Joly F, Vardy J, Ahles T, Dubois M, Tron L, Winocur G, De Ruiter MB, Castel H. Cancer-related cognitive impairment: an update on state of the art, detection, and management strategies in cancer survivors. Ann Oncol. 2019 Dec 1;30(12):1925-1940. doi: 10.1093/annonc/mdz410. PMID 31617564
- [Background] Merzenich MM, Van Vleet TM, Nahum M. Brain plasticity-based therapeutics. Front Hum Neurosci. 2014 Jun 27;8:385. doi: 10.3389/fnhum.2014.00385. eCollection 2014. PMID 25018719
- [Background] Ng EM, Polatajko HJ, Marziali E, Hunt A, Dawson DR. Telerehabilitation for addressing executive dysfunction after traumatic brain injury. Brain Inj. 2013;27(5):548-64. doi: 10.3109/02699052.2013.766927. Epub 2013 Mar 8. PMID 23472964
- [Background] Missiuna C, Mandich AD, Polatajko HJ, Malloy-Miller T. Cognitive orientation to daily occupational performance (CO-OP): part I--theoretical foundations. Phys Occup Ther Pediatr. 2001;20(2-3):69-81. PMID 11345513
- [Background] Wolf TJ, Doherty M, Kallogjeri D, Coalson RS, Nicklaus J, Ma CX, Schlaggar BL, Piccirillo J. The Feasibility of Using Metacognitive Strategy Training to Improve Cognitive Performance and Neural Connectivity in Women with Chemotherapy-Induced Cognitive Impairment. Oncology. 2016;91(3):143-52. doi: 10.1159/000447744. Epub 2016 Jul 23. PMID 27449501
- [Derived] Maeir T, Makranz C, Peretz T, Odem E, Tsabari S, Nahum M, Gilboa Y. Cognitive Retraining and Functional Treatment (CRAFT) for adults with cancer related cognitive impairment: a preliminary efficacy study. Support Care Cancer. 2023 Feb 7;31(3):152. doi: 10.1007/s00520-023-07611-y. PMID 36746805